CLINICAL TRIAL: NCT03055871
Title: Parents and Children Active Together: Examining Motivational, Regulatory, and Habitual Intervention Approaches
Brief Title: Parents and Children Active Together Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 704959
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity
Keywords: Behavioural: Family physical activity habit
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard education control group (No Intervention): The control group package will consist of Canada's PA guidelines recommending 180 min per week for young children, transitioning to 60 minutes of activity a day for children at five and a breakdown of ways for the parent to help their child achieve this PA (unstructured, endurance, strength, activities) commensurate with this guide. The guide also contains arguments and information about the benefits of PA.
- Physical activity planning intervention (Other): The physical activity planning intervention condition will receive the same guidelines as the standard education control group but will also be provided with family physical activity planning material. This material will include workbook on how to plan for family physical activity; brainstorming exercise for children where they list physical activities that they have found fun in the past, as well as activities that they would find enjoyable to do as a family.
  Interventions: Behavioral: Physical activity planning intervention
- Habit formation intervention (Other): The habit formation intervention condition will receive the same content as the education control condition and the physical activity planning condition but with additional material on creating physical activity support habits. The material includes a brief discussion of what habits are with some very straightforward examples such as preparing for sleep routines, or initiating to drive a car to work. A key component of the habit section will be based on planning for context-dependent repetition, with pointers on how to maintain repetition as habit forms.
  Interventions: Behavioral: Habit formation intervention

INTERVENTIONS:
Behavioral: Habit formation intervention — In addition to the control content and the planning content, this intervention will include material provided to the family that assists with creating physical activity support habits. The material contains a discussion of what habits are, straightforward examples, planning and pointers for forming habits. A key component of the habit intervention will be planning for context-dependent repetition.
  Arms: Habit formation intervention
Behavioral: Physical activity planning intervention — This arm will receive the control education content, but will also be provided with family PA planning material. This material will include skill training content (workbook on how to plan for family PA). The material includes a brainstorming exercise for parents where they list physical activities they think their children have found fun in the past, as well as activities that they would find enjoyable to do as a family. We also have Canadian parental survey data on the most preferred co-physical activities for children 3-6. We will provide this material as prompts/suggestions. This list helps create the template for PA planning by contextualizing what the parents would like to do with their kids.
  Arms: Physical activity planning intervention

SUMMARY:
The purpose of this study is to examine physical activity habit formation in parents and if this can increase moderate to vigorous physical activity behavior in their children over six months.The Primary Research Question is:

Does the habit formation condition result in increased moderate-vigorous intensity physical activity of the child compared to the control (education) and education + planning conditions at six months? Hypothesis: Child physical activity will be higher for the habit formation condition in comparison to the more standard physical activity education and planning conditions at six months.

DETAILED DESCRIPTION:
Secondary Research Questions

1. Can group differences among behavioural outcomes be explained through a mediation model? Hypothesis: The covariance of the assigned conditions (habit formation, planning + education, education control) on child PA will be explained by parental co-activity habit, and through the use of consistency and cues regulation strategies (i.e., manipulation check). The habit formation condition will not affect parental support intentions or underlying outcome expectations (benefits of PA) for support of child PA because its effect on behavior is to tie initial intentions to behavioural action or to work independent of goals and intentions.
2. Do factors such as quality of life, parental competence, and family functioning improve with increased PA? Hypothesis: Conditions that increase PA will show commensurate increases in these factors.
3. Is there an intergenerational, seasonal, or gender difference across primary outcomes by assigned condition? Hypothesis: Parents in the habit formation condition will show higher PA via the activities being performed with their children in comparison to the other conditions. No differences in gender or season are hypothesized based on the current research at present

ELIGIBILITY:
Inclusion Criteria:

* Participants will be at least one parent with at least one child between the ages of 3 and 5 years. Families will reside in greater Victoria, British Columbia. Parents can be single parents or co-parents (i.e. we only require one parent and one child to participate). Families will be included if they have at least one parent who will participate and one child between the ages of 3 and 5 who is not meeting current physical activity guidelines (>=60 minutes a day of moderate to vigorous physical activity. There will be no delimitations to the sample based on socio-economic or ethnic variables.

Exclusion Criteria:

* Exclusion Criteria: If child is meeting the current physical activity guidelines >=60 minutes a day of moderate to vigorous physical activity per day.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in children's physical activity to 6 months | Baseline and 6 months
  Children's physical activity will be quantified by accelerometry. Children will wear an accelerometer for a minimum of 6 hours per day for 7 days at baseline and 6 months. Additionally this measure will assess intermediate outcomes at 6 weeks and 3 months.

SECONDARY OUTCOMES:
Change from baseline to 6 months in child physical activity by parent proxy self-report | Baseline and 6 months
  The parent will complete a modified Godin Leisure-Time Exercise Questionnaire to report physical activity of the target child to assess habitual moderate to vigorous physical activity at baseline, 6 weeks, 3 months, 6 months. Questions assess intensity, frequency, and duration of physical activity in an average week. Additionally this measure will assess intermediate outcomes at 6 weeks and 3 months.
Change from baseline in self-reported parental co-activity habit to 6 months | Baseline and 6 months
  The parent will complete an adapted self-reported habit strength index for co-activity with their child at baseline, 6 weeks, 3 months, and 6 months. Intermediate outcomes will be at 6 weeks and 3 months.

OTHER OUTCOMES:
TERTIARY OUTCOME - Change from baseline in parent physical activity to 6 months | Baseline and 6 months
  Parental physical activity will be quantified by accelerometry. Parents will wear an accelerometer for a minimum of 10 hours per day for 7 days at baseline and 6 months. Additionally this measure will assess intermediate outcomes at 6 weeks and 3 months.
TERTIARY OUTCOME - Change from baseline to 6 months in self-reported parent physical activity | Baseline and 6 months
  As a tertiary outcome measure, the Godin Leisure-Time Exercise Questionnaire will be used to measure self-reported physical activity at baseline, 6 weeks, 3 months, 6 months. Questions assess intensity, frequency, and duration of physical activity in an average week.
TERTIARY OUTCOME - Change from baseline in self-reported parent-child co-activity to 6 months | Baseline and 6 months
  Parents will complete a modified Godin Leisure Time Exercise Questionnaire to assess parent-child co-activity. This measure will be assessed at baseline, 6 weeks, 3 months, and 6 months. Intermediate outcomes will be at 6 weeks and 3 months.
TERTIARY OUTCOME - Change from baseline in objectively assessed parent-child co-activity to 6 months. | Baseline and 6 months
  An accelerometer Bluetooth-enabled feature measures proximity detection, allowing for the objective assessment of co-activity between parent and child. Parent and child will wear accelerometers at baseline, 6 weeks, 3 months, and 6 months to assess co-activity. Intermediate co-activity outcomes will be at 6 weeks and 3 months.
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 6 weeks | Baseline and 6 weeks
  Tertiary Outcome Measure Motivations for parent-child co-activity will be measured using affective attitude, instrumental attitude, perceived capability, behavioural regulation, intention, automaticity and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 3 months | Baseline and 3 months
  Tertiary Outcome Measure Motivations for parent-child co-activity will be measured using affective attitude, instrumental attitude, perceived capability, behavioural regulation, intention, automaticity and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
TERTIARY OUTCOME - Change from baseline in motivations (MPAC constructs) at 6 months | Baseline and 6 months
  Tertiary Outcome Measure Motivations for parent-child co-activity will be measured using affective attitude, instrumental attitude, perceived capability, behavioural regulation, intention, automaticity and identity. These measures are all part of the Multi Process Action Control Framework (MPAC).
TERTIARY OUTCOME - Change from baseline in health-related quality of life at 6 months | Baseline and 6 months
  Tertiary Outcome Measure Quality of life will be assessed with parents using the 12 item Short Form Health Survey. Change in health-related quality of life from baseline to 6 months (i.e., post-intervention) will be examined with intermediate time points of 6 weeks and 3 months as well.
TERTIARY OUTCOME - Change from baseline in parental competence at 6 months | Baseline and 6 months
  Tertiary Outcome Measure Parental competence will be measured via the Parenting Sense of Competence Scale at baseline and 6 months with intermediate time points of 6 weeks and 3 months.
TERTIARY OUTCOME - Change from baseline in family functioning at 6 months | Baseline and 6 months
  Tertiary Outcome Measure Family Environment Scale is used to assess family functioning at baseline, 6 weeks, 3 months, and 6 months.
MANIPULATION CHECK - Change from baseline to 6 months in cue consistency | Baseline and 6 months
  To examine the manipulation check outcomes, a 6 item survey assessing the utilization of context-dependent repetition/cues and consistency/repeated action is used. Changes in cue consistency will be examined at 6 months with intermediate time points of 6 weeks and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Mark Beauchamp, PhD, Study Chair — University of British Columbia; Chris Blanchard, PhD, Study Chair — Dalhousie University; Valerie Carson, PhD, Study Chair — University of Alberta; Benjamin Gardner, PhD, Study Chair — King's College; Darren Warburton, PhD, Study Chair — University of British Columbia
Locations (1):
- Behavioural Medicine Lab, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grant SJ, Beauchamp MR, Blanchard CM, Carson V, Gardner B, Warburton DER, Rhodes RE. Parents and children active together: a randomized trial protocol examining motivational, regulatory, and habitual intervention approaches. BMC Public Health. 2020 Sep 21;20(1):1436. doi: 10.1186/s12889-020-09465-z. PMID 32957959